CLINICAL TRIAL: NCT05558072
Title: Is There a Toll-like 4 Receptor Relationship in Patients With Testicular Torsion?
Brief Title: Testicular Torsion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hisar Intercontinental Hospital (Other)
Responsible Party: Principal Investigator, Basri Cakiroglu, Ass. Prof., Hisar Intercontinental Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2022/18
Record Dates: First submitted 2022-09-23; First posted 2022-09-28 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Testicular Torsion and TLR 4 Was Investigated
Keywords: testicular torsion,; Toll-like receptors (TLR),; child; newborn; adolescent
MeSH Terms: conditions — Spermatic Cord Torsion | interventions — Toll-Like Receptor 4

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Newborn
  Interventions: Genetic: Toll-like receptor 4
- Group 2 (Experimental): adolescent
  Interventions: Genetic: Toll-like receptor 4

INTERVENTIONS:
Genetic: Toll-like receptor 4 — Toll-like receptor 4

SUMMARY:
Background:

Testicular torsion is a scrotal emergency that results in impaired blood supply to the testis and ischemia of the testis as a result of the rotation of the spermatic cord around itself. The etiology of testicular torsion is not clear, but various predisposing factors are responsible for the occurrence of testicular torsion.

Recently, with the discovery of "Toll-Like Receptors" (TLRs), new horizons have been opened in the field of innate immune system-related diseases.

Objective: To mediate the relationship between testicular torsion and TLR4 receptors.

Material-Method: Testicular specimens of patients who developed testicular ischemia after testicular torsion and underwent orchiectomy between 2012-2022 were reached. A study of TLR 4 receptors was performed in these testicular specimens. The patients were divided into two groups according to their ages newborns and adolescents.

DETAILED DESCRIPTION:
Analysis of 32 newborns and 32 adolescents between the ages of 14 and 16 (mean age was 15.17 ± 0.98) testicular tissue lysate using Toll-Like Receptor antibody 4 (TLR4) ELISA (Enzyme-Linked ImmunoSorbent Assay).

Toll-like receptor 4 is a transmembrane protein that in humans is encoded by the TLR4 gene. Its activation leads to the production of inflammatory cytokines.

ELIGIBILITY:
Inclusion Criteria:

testicular torsion

* newborn, adolescent,

Exclusion Criteria:

* orchitis, urinary infection, trauma,

Ages: 0 Days to 16 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — Testis torsion
Enrollment: 64 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Toll-like receptor 4 positives or negative | 10 years
  testicular torsion

IPD SHARING:
Plan to Share IPD: No